CLINICAL TRIAL: NCT00993265
Title: Double-Blind, Placebo-Controlled Trial of N-acetylcysteine for the Treatment of Pediatric Trichotillomania
Brief Title: N-Acetylcysteine for Pediatric Trichotillomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Trichotillomania Learning Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0906005337; NACPEDTTM
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Trichotillomania; Hair Pulling
Keywords: Trichotillomania; Hair pulling; glutamate; N-Acetylcysteine; Children
MeSH Terms: conditions — Trichotillomania | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (NAC) (Experimental): Patients randomized to this arm will receive N-Acetylcysteine, at a standard dose titrated to 2400 mg. They will receive NAC in addition to the medication regimen they are on at enrollment.
  Interventions: Drug: N-Acetylcysteine
- Placebo (Placebo Comparator): Patients randomized to this arm will receive placebo, formulated to be indistinguishable from N-Acetylcysteine, in addition to the medication regimen they are on at study enrollment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — 2400 mg by mouth PO (1200 mg AM, 1200 mg PM), 12 weeks
  Arms: N-acetylcysteine (NAC)
Drug: Placebo — placebo, 2 capsules by mouth in AM, 2 capsules by mouth PM, 12 weeks
  Arms: Placebo

SUMMARY:
Trichotillomania (hair pulling) has an estimated lifetime prevalence of 1-3%. Children with trichotillomania can experience significant impairment due to peer teasing, avoidance of activities (such as swimming and socializing), difficulty concentrating on school work and medical complications due to pulling behaviors. Despite the fact that trichotillomania has a childhood onset, no randomized, controlled trials have been completed in childhood trichotillomania.

Research in adults with trichotillomania has demonstrated that most commonly currently prescribed treatment for trichotillomania, (pharmacotherapy with selective serotonin reuptake inhibitors) is ineffective in treating this condition. By contrast, randomized controlled trials in adults have suggested the efficacy of N-acetylcysteine as well as behavioral treatments such as Habit Reversal Therapy.

The goal of this trial is to determine the efficacy of N-Acetylcysteine for pediatric trichotillomania. N-Acetylcysteine is a glutamate modulating agent, with a fairly benign side-effect profile.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-17 years.
* Primary DSM-IV diagnosis of trichotillomania or chronic hair pulling.
* Duration of trichotillomania greater than 6 months.

Exclusion Criteria:

* Comorbid bipolar disorder, psychotic disorder, substance use disorder, developmental disorder or mental retardation (IQ<70).
* Recent change (less than 4 weeks) in medications that have potential effects on TTM severity (such as SSRIs, CMI, naltrexone, lithium, psychostimulants, anxiolytics, or antipsychotics). Medication change is defined to include either dose changes or medication discontinuation.
* Asthma requiring medication use within the last 6 months.
* Known hypersensitivity or previous anaphylactoid reaction to acetylcysteine or any components in its preparation
* Current use (within last week) of psychostimulant medications.
* Positive pregnancy test or drug screening test

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, M.D., M.S., Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Bloch MH. Trichotillomania across the life span. J Am Acad Child Adolesc Psychiatry. 2009 Sep;48(9):879-883. doi: 10.1097/CHI.0b013e3181ae09f3. No abstract available. PMID 19692854
- [Background] Grant JE, Odlaug BL, Kim SW. N-acetylcysteine, a glutamate modulator, in the treatment of trichotillomania: a double-blind, placebo-controlled study. Arch Gen Psychiatry. 2009 Jul;66(7):756-63. doi: 10.1001/archgenpsychiatry.2009.60. PMID 19581567
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562
- [Derived] Schumer MC, Panza KE, Mulqueen JM, Jakubovski E, Bloch MH. LONG-TERM OUTCOME IN PEDIATRIC TRICHOTILLOMANIA. Depress Anxiety. 2015 Oct;32(10):737-43. doi: 10.1002/da.22390. Epub 2015 Jul 2. PMID 26139231
- [Derived] Panza KE, Pittenger C, Bloch MH. Age and gender correlates of pulling in pediatric trichotillomania. J Am Acad Child Adolesc Psychiatry. 2013 Mar;52(3):241-9. doi: 10.1016/j.jaac.2012.12.019. PMID 23452681
- [Derived] Bloch MH, Panza KE, Grant JE, Pittenger C, Leckman JF. N-Acetylcysteine in the treatment of pediatric trichotillomania: a randomized, double-blind, placebo-controlled add-on trial. J Am Acad Child Adolesc Psychiatry. 2013 Mar;52(3):231-40. doi: 10.1016/j.jaac.2012.12.020. PMID 23452680

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine (NAC) | Placebo
Started | 20 | 19
Completed | 16 | 19
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Changed dose of concomitant drug | 2 | 0
Not completed — Non-compliant with study medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine (NAC) | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 19 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (2.4) | 13.1 (3.1) | 13.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39
Massachusetts General Hospital - Hairpulling Scale (MGH-HPS) [Mean (Standard Deviation); unit: units on a scale] — The Massachusetts General Hospital - Hairpulling Scale (MGH-HPS) is a 7-question scale that measures the severity of hair pulling. The scale ranges from 0-28. The higher the score, the more severe the hairpulling.
  units on a scale | 13.2 (5.3) | 16.6 (4.8) | 14.9 (5.3)
The Trichotillomania Scale for Children (TSC)-Child Report [Mean (Standard Deviation); unit: units on a scale] — The Trichotillomania Scale for Children (TSC) - Child Version assesses hair pulling severity, distress, and impairment in children. The scale is split into two sections (severity and distress/impairment), with 12 questions (5 severity and 7 distress/impairment). The severity score is summed from questions 1-5 and divided by 5. The distress/impairment score is summed from questions 6-12 and divided by 7. The total score is calculated by summing the severity score and the distress/impairment score. Scores range from 0-4. Higher total scores indicate greater severity/distress/impairment.
  units on a scale | 2.35 (.74) | 2.52 (.85) | 2.44 (.85)
The Trichotillomania Scale for Children (TSC)-Parent Report [Mean (Standard Deviation); unit: units on a scale] — The Trichotillomania Scale for Children (TSC) - Parent Version assesses hair pulling severity, distress, and impairment in children. The scale is split into two sections (severity and distress/impairment), with 12 questions (5 severity and 7 distress/impairment). The severity score is summed from questions 1-5 and divided by 5. The distress/impairment score is summed from questions 6-12 and divided by 7. The total score is calculated by summing the severity score and the distress/impairment score. Scores range from 0-4. Higher total scores indicate greater severity/distress/impairment.
  units on a scale | 2.20 (0.71) | 2.32 (0.71) | 2.26 (0.71)
The Milwaukee Inventory for Styles of Trichotillomania (MIST) - Child Version [Mean (Standard Deviation); unit: units on a scale] — The Milwaukee Inventory for Styles of Trichotillomania (MIST) - Child Version assesses "focused" pulling, hair pulling that occurs intentionally to relieve tension or distress, and "automatic" pulling, hair pulling that occurs outside of the child's attention. This scale contains 25 questions, 21 questions in the "focused" pulling subscale and 4 questions in the "automatic" pulling subscale. The scores range from 0-36 on the "automatic" pulling subscale and 0-189 on the "focused" pulling subscale. Higher scores on the subscales indicate more of the hair pulling is of that style.
  units on a scale
    Baseline MIST-C Focused Pulling Subscale | 94 (35.2) | 90.8 (30.5) | 92.4 (35.2)
    Baseline MIST-C Automatic Pulling Subscale | 12.10 (9.3) | 16.26 (9.8) | 14.18 (9.8)
Multidimensional Anxiety Scale for Children (MASC) [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Anxiety Scale for Children (MASC) assesses major dimensions of anxiety in children. The MASC contains 39 items rated on a scale of 0-3. Scores range from 0-117. The higher the score, the greater the anxiety.
  units on a scale | 48.7 (19.0) | 52.9 (18.6) | 50.8 (19.0)
The Children's Depression Inventory (CDI) [Mean (Standard Deviation); unit: units on a scale] — The Children's Depression Inventory (CDI) assesses depressive symptoms in children. The assessment contains 27 items rated on a scale of 0-2, with scores ranging from 0-54. The higher the score, the more severe the depressive symptoms.
  units on a scale | 12.4 (6.8) | 10.8 (8.5) | 11.6 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Massachusetts General Hospital Hair Pulling Scale (MGH-HPS)
Description: The Massachusetts General Hospital - Hairpulling Scale (MGH-HPS) is a 7-question scale that measures the severity of hair pulling. The scale ranges from 0-28. The higher the score, the more severe the hairpulling.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 20 | 19
units on a scale | 10.70 (1.49) | 13.53 (1.47)

2. Secondary Outcome: Trichotillomania Scale for Children - Child Version
Description: The Trichotillomania Scale for Children (TSC) - Child Version assesses hair pulling severity, distress, and impairment in children. The scale is split into two sections (severity and distress/impairment), with 12 questions (5 severity and 7 distress/impairment). The severity score is summed from questions 1-5 and divided by 5. The distress/impairment score is summed from questions 6-12 and divided by 7. The total score is calculated by summing the severity score and the distress/impairment score. Scores range from 0-4. Higher total scores indicate greater severity/distress/impairment.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 20 | 19
units on a scale | 2.00 (0.22) | 2.08 (0.22)

3. Secondary Outcome: Multidimensional Anxiety Scale for Children (MASC)
Description: The Multidimensional Anxiety Scale for Children (MASC) assesses major dimensions of anxiety in children. The MASC contains 39 items rated on a scale of 0-3. Scores range from 0-117. The higher the score, the greater the anxiety.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 20 | 19
units on a scale | 48.4 (4.3) | 49.8 (4.3)

4. Secondary Outcome: Children's Depression Inventory
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 20 | 19
units on a scale | 10.9 (1.9) | 7.8 (1.9)

5. Secondary Outcome: Trichotillomania Scale for Children - Parent Version
Description: The Trichotillomania Scale for Children (TSC) - Parent Version assesses hair pulling severity, distress, and impairment in children. The scale is split into two sections (severity and distress/impairment), with 12 questions (5 severity and 7 distress/impairment). The severity score is summed from questions 1-5 and divided by 5. The distress/impairment score is summed from questions 6-12 and divided by 7. The total score is calculated by summing the severity score and the distress/impairment score. Scores range from 0-4. Higher total scores indicate greater severity/distress/impairment.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 20 | 19
units on a scale | 1.83 (0.18) | 1.88 (0.18)

6. Secondary Outcome: The Milwaukee Inventory for Styles of Trichotillomania-Child Version
Description: The Milwaukee Inventory for Styles of Trichotillomania (MIST) - Child Version assesses "focused" pulling, hair pulling that occurs intentionally to relieve tension or distress, and "automatic" pulling, hair pulling that occurs outside of the child's attention. This scale contains 25 questions, 21 questions in the "focused" pulling subscale and 4 questions in the "automatic" pulling subscale. The scores range from 0-36 on the "automatic" pulling subscale and 0-189 on the "focused" pulling subscale. Higher scores on the subscales indicate more of the hair pulling is of that style.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 20 | 19
units on a scale
  Week 12 MIST-C "Automatic" Subscale | 13.24 (1.98) | 13.16 (1.96)
  Week 12 MIST-C "Focused" Subscale | 90.8 (8.1) | 79.6 (8.1)

7. Secondary Outcome: National Institute of Mental Health -Trichotillomania Severity Scale (NIMH-TSS)
Description: The National Institute of Mental Health - Trichotillomania Severity Scale (NIMH-TSS) assesses severity of hair pulling. The NIMH-TSS is a 6 item assessment, with total scores ranging from 0-20. Higher scores indicate greater severity/impairment.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 20 | 19
units on a scale | 9.56 (0.71) | 10.89 (1.24)

ADVERSE EVENTS:
Arm/Group | N-acetylcysteine (NAC) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 6/20 | 12/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine (NAC) (N=20) | Placebo (N=19)
Nausea (Gastrointestinal disorders) | 6 | 12
Diarrhea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Insomnia (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Difficulty Swallowing Pills (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes